CLINICAL TRIAL: NCT02579083
Title: A Phase 1, Single Center Study to Assess the Safety of MB66, a Combined Anti-HIV (VRC01-N) and Anti-HSV (HSV8-N) Monoclonal Antibody Film for Vaginal Application as Microbicide
Brief Title: Safety Study of Monoclonal Antibodies to Reduce the Vaginal Transmission of HSV and HIV
Acronym: VAST
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KBio Inc (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Boston University (Other); The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MB66-01; U19AI096398 (NIH)
Record Dates: First submitted 2015-10-09; First posted 2015-10-19 (Estimated); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: HIV; Herpes Simplex Infections
MeSH Terms: conditions — Herpes Simplex

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Segment A: Single MB66 Administration (Experimental): 10 mg of HSV8-N and 10 mg of VRC01-N monoclonal antibodies per MB66 film
  Interventions: Drug: MB66
- Segment B: Repeated Administrations Placebo Film (Placebo Comparator): The placebo film is composed of the identical excipients as MB66 without the monoclonal antibodies.
  Interventions: Drug: Placebo Film
- Segment B: Repeated Administrations MB66 (Experimental): 10 mg of HSV8-N and 10 mg of VRC01-N monoclonal antibodies per MB66 film
  Interventions: Drug: MB66

INTERVENTIONS:
Drug: MB66 — 10 mg of HSV8-N and 10 mg of VRC01-N monoclonal antibodies per MB66 film
  Other Names: Investigational Product
  Arms: Segment A: Single MB66 Administration; Segment B: Repeated Administrations MB66
Drug: Placebo Film — The placebo film is composed of the identical excipients as MB66 without the monoclonal antibodies.
  Other Names: Placebo
  Arms: Segment B: Repeated Administrations Placebo Film

SUMMARY:
The purpose of this study is to assess the safety and pharmacokinetics of MB66, a monoclonal antibody film for vaginal application that is being developed to potentially reduce the transmission of herpes simplex virus (HSV) and human immunodeficiency virus (HIV).

DETAILED DESCRIPTION:
This is a single center, Phase 1, randomized, single blind, placebo-controlled, two-segment study to assess the safety of the MB66 vaginal film. After appropriate screening, approximately 43 healthy women will be enrolled. The study will be divided into two sequential Segments. The first, Segment A, is a single-arm, single-dose, open label design. The 8 Segment A participants will receive a single dose of one full MB66 film. After dosing, subjects will be asked to maintain sexual abstinence and will be evaluated in person on Day 1 (24-hours post MB66 administration), by telephone on Day 3 or 4 and in person on the Day 6-10 Exit Visit, after which subjects will be allowed to resume sexual activity with study-provided condoms until three weeks after last exposure to film (to avoid male exposure to residual drug product). A placebo arm is not included in Segment A, because the very low risk of toxicity of the placebo film makes it unlikely that any toxicity observed in Segment A would be wrongly attributed to the active agents (mAbs) in the MB66 film. This conclusion is based on the known tolerance of the very similar vehicle used in a commercial polyvinyl alcohol (PVA)-based vaginal film (VCF®), and the absence of toxicity of the MB66 placebo film in the very sensitive rabbit model after substantially higher dosing intensity and duration.

Completion of Segment A and a safety review of Segment A adverse events will trigger the initiation of Segment B, a repeat dose, randomized, two arm, single-blind, placebo-controlled design. Subjects will be randomized 1:1 into two groups (15 evaluable subjects per group) and be treated once daily with either 1 MB66 film or 1 vehicle control placebo film for seven consecutive days. For five days before, and for 7 days after the dosing period, subjects will be asked to maintain a period of sexual abstinence. Subjects will be evaluated in person on Day 0 (at 1 and 4 hours post MB66 in-clinic dosing), again on Day 1 (24 hr post dosing), by telephone on Day 3-4, and evaluated again in person on Day 7-8, after which, subjects will be allowed to resumed sexual activity with condoms required until three weeks after last film insertion. Subjects will be evaluated a last time on the Day 12-16 Exit Visit.

In addition to safety measures, pharmacokinetic evaluations will be done on Day 0, Day 1, and Day 7 in both Segments, and additionally on Day 14 for Segment B. Specifically, this study will evaluate the rate of MB66 film dissolution, the vaginal concentrations of the MB66 antibodies, and the degree of systemic absorption of the MB66 antibodies. A number of of exploratory objectives will also be evaluated, including assessment of the antiviral effect of the MB66 antibodies ex vivo in cervicovaginal lavage fluid from participants after dosing with MB66 film, the effects of MB66 and placebo films on the cervicovaginal microbial environment using pH, Nugent score, and bacterial ribosomal DNA polymerase chain reaction (PCR), and comparison of the effect of MB66 and placebo films on cervicovaginal immune mediators by Luminex and ELISA assays. Segment B participants will also be asked to assess the acceptability of the MB66 vaginal film after 7 days of use.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 through 45 years (inclusive) at screening
2. Able and willing to provide written informed consent to be screened for and enrolled in the study
3. Able and willing to provide adequate locator information at screening
4. HIV-uninfected based on testing performed by study staff at
5. In general good health as determined by the site clinician
6. Agree to abstain from any vaginal insertions, including products, douches, devices such as sex toys, or penile or oral intercourse from 5 days prior to Visit 2 (Enrollment Visit) until the final Study Visit (one week after last dose of study film). Only tampons during menses and clinically indicated speculum exams are allowed.
7. Agree to use condoms provided by the study staff from one week after last use of study film until three weeks after last use of study film
8. Willingness to undergo all study-related assessments and follow all study-related procedures
9. Be currently using an effective method of contraception at enrollment (used continuously and with good compliance for the past 60 days as determined by participant self-report) with plans to continue use throughout the study period. Acceptable methods include any hormonal method (except vaginal ring); intrauterine device (IUD) inserted at least 90 days prior to enrollment; female sterilization; abstinent from sexual activity with male partner for the past 60 days; sexual activity with vasectomized partner; engages in sex exclusively with women.
10. For participants 21 and older, a Pap result in the 36 calendar months prior to the Enrollment Visit consistent with Grade 0 according to the Female Genital Grading Table for Use in Microbicide Studies Addendum 1 to the DAIDS Table for Grading Adult and Pediatric Adverse Events satisfactory evaluation with no treatment required of non-Grade 0 Pap result per American Society for Colposcopy and Cervical Pathology (ASCCP) guidelines or per local standard of care, within the last 36 calendar months prior to enrollment. Note: For participants aged 18-21, a Grade-0 or adequately evaluated abnormal Pap smear is not required as the American Society for Colposcopy and Cervical Pathology recommends initiating screening at age 21.
11. At screening and enrollment, agrees not to participate in other research studies involving drugs, medical devices, or vaginal products while enrolled in this trial -

Exclusion Criteria:

1. Menopausal at screening (as defined as amenorrhea or irregular periods for one year or more without an alternative etiology)
2. Hysterectomy
3. Known adverse reaction to any of the study products (ever)
4. Known adverse reaction to latex (ever)
5. Non-therapeutic injection drug use in the 12 months prior to screening
6. Surgical procedure involving the pelvis in the 90 days prior to screening (includes dilation and curettage or evacuation, and cryosurgery; does not include cervical biopsy for evaluation of an abnormal pap smear or IUD placement)
7. Participation in a drug, spermicide and/or microbicide study in the 30 days prior to screening or anticipated participation in an investigational drug study in the next 8 weeks
8. Pregnancy within 90 days prior to screening
9. Lactating
10. Use of a diaphragm, NuvaRing®, or spermicide for contraception
11. As determined by the PI, a degree of menstrual cycle irregularity that would make it difficult to schedule follow up visits without interruption by menses
12. Active sexually transmitted infection or documented treatment of sexually transmitted infections in the last 6 months, including, but not limited to: chlamydia, gonorrhea, syphilis, trichomonas, cervicitis or pelvic inflammatory disease, or currently active HSV lesions or other sores. (Participants seropositive for or with a history of HSV without current active lesions will not be excluded.)
13. Women who by history engage in condom-less intercourse with HIV-infected partners, or who exchange sex for money, shelter, or gifts, or who in the opinion of the investigators, may be at risk for HIV acquisition during the duration of the study
14. More than one sex partner within the past 3 months
15. Current sexual partner known by participant to be HIV seropositive
16. Current or planned use of pre-exposure prophylaxis against HIV infection
17. Currently active genital HSV lesions, or other genital tract epithelial disruption or inflammation
18. Current or episodic use of anti-herpes suppressive therapy
19. Urinary tract infection, symptomatic candidiasis, or symptomatic bacterial vaginosis within 14 days of enrollment, or currently residual symptoms thereof Note: women with these infections at screening can be enrolled after treatment and resolution of the infection.
20. Antibiotic or antifungal therapy (vaginal or systemic) within 7 days of enrollment
21. Use of systemic immunomodulatory medications within 4 weeks of enrollment
22. Menses or other vaginal bleeding at the time of enrollment* or expecting menses in the 10 days after enrollment (Segment A participants) or 16 days after enrollment (for Segment B participants)

    *Note: for women with monthly cycles, every attempt will be made to enroll these participants in the first half of their menstrual cycle. Women who have vaginal bleeding at the scheduled Enrollment Visit may return at a different date to be re-examined and possibly enrolled provided they are still within the screening window and meet all criteria.
23. Lack of stable living conditions to allow reliable room temperature storage of study product (Segment B participants only)
24. At enrollment has any of the following laboratory abnormalities per the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.0, Nov 2014:

    * Grade 1 or higher AST (aspartate aminotransferase) or ALT (alanine aminotransferase)
    * Grade 1 or higher creatinine
    * Grade 2 or higher hemoglobin
    * Grade 1 or higher platelets Note: otherwise eligible participants with an exclusionary test may be re-tested once during the screening process.
25. As determined by the Principal Investigator (PI), any subject who has any significant uncontrolled active or chronic cardiovascular, renal, liver, hematologic, neurologic, gastrointestinal, psychiatric, endocrine, respiratory, immunologic disorder or infectious disease, anticoagulation with warfarin or heparin; or any other condition that, in the opinion of the Investigator, would preclude provision of consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2016-01; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Incidence of Grade 2 or higher Adverse Events deemed related to study product | Segment A, cumulative events to Day 7; Segment B, cumulative events to Day 10
  Grade 2 or higher Adverse Events

SECONDARY OUTCOMES:
Naked eye visual assessment during speculum exam of the degree of film dissolution | 1, 4, and 24 hours after dosing
  visual assessment during speculum exam
Concentrations of MB66 antibodies in vaginal fluid sampled with Tear Flo (filter paper) wicks, and measured by enzyme linked immunosorbent assay (ELISA) | Pre-dose, 1 hr and 4 hr post dose, day 1, day 6-10 and day 12-16 (Segment B only)
  Concentrations of MB66 antibodies in vaginal fluid
Concentrations of MB66 antibodies in serum by ELISA | Screening visit, day 1, day 6-10 and day 12-16 (segment B only)
  Concentrations of MB66 antibodies in serum

CONTACTS AND LOCATIONS:
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Politch JA, Cu-Uvin S, Moench TR, Tashima KT, Marathe JG, Guthrie KM, Cabral H, Nyhuis T, Brennan M, Zeitlin L, Spiegel HML, Mayer KH, Whaley KJ, Anderson DJ. Safety, acceptability, and pharmacokinetics of a monoclonal antibody-based vaginal multipurpose prevention film (MB66): A Phase I randomized trial. PLoS Med. 2021 Feb 3;18(2):e1003495. doi: 10.1371/journal.pmed.1003495. eCollection 2021 Feb. PMID 33534791